CLINICAL TRIAL: NCT03321604
Title: Kidney Information Network for Disease Research and Education (KINDRED)
Brief Title: Kidney Information Network for Disease Research and Education
Acronym: KINDRED
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Scott and White Hospital & Clinic (Other)
Responsible Party: Principal Investigator, Ravi Thadhani, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2016P002671
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: ESRD; Fabry Disease; Rare Diseases; Kidney Diseases; End Stage Renal Disease; Genetic Diseases, X-Linked
Keywords: Hemodialysis; Kidney; Dialysis; Kindred; Fabry; Massachusetts General Hospital
MeSH Terms: conditions — Kidney Failure, Chronic; Fabry Disease; Rare Diseases; Kidney Diseases; Genetic Diseases, X-Linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, Investigators will conduct a prospective cohort study of dialysis patients by collecting research-quality information on patient characteristics, comorbid diseases and laboratory markers used in routine practice, as well as novel biochemical markers and genetic data. Investigators will utilize data from the cohort to test the independent relationship between biochemical and genetic markers and Fabry disease and other rare diseases.

DETAILED DESCRIPTION:
KINDRED is a prospective observational cohort study that will enroll up to 5,000 dialysis patients throughout the United States with and without known diagnosis of Fabry disease but at risk for Fabry disease (e.g., unknown cause of renal disease, young male, initiating dialysis without a kidney biopsy, etc).This tissue repository will allow for genetic screening of a geographically diverse population, assist in identification of rare diseases in ESRD, and collect research-quality information on risk factors and outcomes from an ethnically heterogeneous population of dialysis patients. In this study, Investigators will use a novel method of performing research in this population by leveraging the internet to enhance and accelerate recruitment of potential subjects to participate in a genetic screening/tissue repository protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 with ESRD undergoing dialysis.

Exclusion Criteria:

* Kidney biopsy unlikely to be Fabry disease; those with a diagnosis that is clinically or biochemically proven not to be Fabry disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving dialysis
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Genetically determined Fabry disease prevalence amongst a heterogenous patient population with end-stage renal disease on dialysis in the US not previously known to have Fabry disease. | 5 years

SECONDARY OUTCOMES:
Differences in patient characteristics of dialysis patients diagnosed with Fabry disease vs. dialysis patients who do not have Fabry disease. | 5 years
Differences in patient characteristics of individuals diagnosed with Fabry disease initiating dialysis after 2013 vs. patients with Fabry disease who started dialysis before 2003. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: KINDRED Website — https://kindredresearch.mgh.harvard.edu